CLINICAL TRIAL: NCT05166928
Title: Effect of Upper Third Molar Extraction on Distalization Using Carriere Motion Appliance :A Prospective Clinical Study
Brief Title: Effect of Upper Third Molar Extraction on Distalization Carriere Motion Appliance :A Prospective Clinical Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Nassem mohsen qasem, faculty of dental medicine (Cairo-boys) AL-Azhar University, Al-Azhar University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 627/1151
Record Dates: First submitted 2021-12-12; First posted 2021-12-22 (Actual); Last update posted 2021-12-22 (Actual); Status verified 2021-12

CONDITIONS: Class II Malocclusion
MeSH Terms: conditions — Overbite

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1: control group (Active Comparator): will be treated using carriere motion appliance for distalization of upper buccal segment in the presence of upper third molar
  Interventions: Device: carriere motion appliance
- group2: teste group (Active Comparator): will be treated with using carriere motion appliance for distalization of upper buccal segment with upper third molar extraction or have congenital missing upper third molar
  Interventions: Device: carriere motion appliance

INTERVENTIONS:
Device: carriere motion appliance — after finished treatment with carrirere motion appliance in the two group (group 1 have upper wisdom teeth ,group 2 have not upper wisdom teeth ) the pre and post casts will be scanned and superimposed to determine amount upper molar distalization

SUMMARY:
This clinical study will be directed to compare the effect of presence or absence of third molar on distalization of the upper posterior segment by using carriere motion appliance

ELIGIBILITY:
Inclusion Criteria:

1. Angle´s Class II canine relationship, at least half-unit.
2. Skeletal Class I or mild Class II relationship.
3. Upper second molars were fully erupted before starting distalization.
4. Normal or horizontal growth pattern.
5. Good oral hygiene.
6. Absence of any systemic diseases

Exclusion Criteria:

Previous orthodontic treatment. 2. Patients who required surgery to correct skeletal discrepancies (sever skeletal class11).

3. Patients with hyperdontia, hypodontia, or syndromic diseases. 4. Extraction or badly destructed teeth in upper arch

-

Ages: 14 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2021-07-10 (Actual); Primary Completion 2021-11-10 (Actual); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
change in upper first molar position | Baseline to 6 months
  using 3d cast superimposition

CONTACTS AND LOCATIONS:
Locations (1):
- al-Azhar university, Cairo, Naser Ciry, Egypt

IPD SHARING:
Plan to Share IPD: Undecided